CLINICAL TRIAL: NCT00177333
Title: Serum Levels of Doxycycline at the Time of Abortion With Two Dosing Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: pittirb0504092
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Abortion, Induced; Vomiting
Keywords: Abortion, Induced; Doxycycline; Antibiotic Prophylaxis; Vomiting; Abortion, Therapeutic
MeSH Terms: conditions — Vomiting | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Doxycycline

SUMMARY:
This is a randomized double-blind, controlled trial comparing two regimens of pre-abortion doxycycline. The aims of the study are to determine the serum levels of doxycycline when administered pre-operatively 4 hours or approximately 18 hours before a dilation and evacuation (D & E) abortion. The hypotheses being tested are that subjects who receive doxycycline with food the night before an abortion will have adequate serum levels, but less nausea and vomiting compared to women who take the doxycycline on an empty stomach on the morning of the abortion. Subjects will either take 200mg doxycycline on the night before and 2 caps placebo with a sip of water on the morning of surgery or 2 caps placebo the night before and 200mg doxycycline on the morning of surgery with a sip of water. All capsules will look identical. Diaries, questionnaires and a 10cc sample of blood for doxycycline levels will be collected from the subjects at the time of surgery.

DETAILED DESCRIPTION:
This is a randomized double-blind, controlled trial comparing two regimens of pre-abortion doxycycline. The aims of the study are to determine the serum levels of doxycycline when administered pre-operatively 4 hours or approximately 18 hours before a dilation and evacuation (D & E) abortion. The hypotheses being tested are that subjects who receive doxycycline with food the night before an abortion will have adequate serum levels, but less nausea and vomiting compared to women who take the doxycycline on an empty stomach on the morning of the abortion. Subjects will either take 200mg doxycycline on the night before and 2 caps placebo with a sip of water on the morning of surgery or 2 caps placebo the night before and 200mg doxycycline on the morning of surgery with a sip of water. All capsules will look identical. Diaries, questionnaires and a 10cc sample of blood for doxycycline levels will be collected from the subjects at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 15-23 weeks by ultrasound.
2. Willing and able to sign an informed consent.
3. Placement of cervical dilators. Dilators must be placed before giving any subject doxycycline in order to ensure that all subjects who receive doxycycline will have an abortion.
4. Willing to comply with the study protocol.
5. Age at enrollment of 18 years or more.

Exclusion Criteria:

1. Need for an urgent D & E. Indications for this include ruptured membranes, advanced cervical dilation, infection, and fetal demise.
2. Allergy to doxycycline or any tetracycline
3. Exposure to or treatment for gonorrhea or chlamydia within the past 90 days.
4. Current or recent (within the past week) use of any other antibiotic.
5. Prior cardiac valve surgery or cardiac valve replacement. These patients should all receive alternative antibiotics for endocarditis prophylaxis.
6. Active use of alcohol, heroin, or cocaine. Active use of alcohol will be defined as more than 2 drinks per day. Any use of heroin or cocaine will be considered exclusionary.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
doxycycline side effects | 24 hours

SECONDARY OUTCOMES:
nausea | 24 hours
vomiting | 24 hours
other side effects | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: M Reeves, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Reeves MF, Lohr PA, Harwood BJ, Creinin MD. Ultrasonographic endometrial thickness after medical and surgical management of early pregnancy failure. Obstet Gynecol. 2008 Jan;111(1):106-12. doi: 10.1097/01.AOG.0000296655.26362.6d. PMID 18165398